CLINICAL TRIAL: NCT06586749
Title: The Effect of Patient Education and Implementation of Teleinterventions by Nurses, on the Incidence of Surgical Wound Infections, in Patients After Coronary Artery Bypass Surgery
Brief Title: Effect of Nurse-Led Education and Tele-Interventions on Reducing Surgical Site Infections in Patients After Coronary Artery Bypass Surgery: a Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Mediterranean University (Other)
Responsible Party: Principal Investigator, Konstantinos Giakoumidakis, Associate Professor, Department of Nursing, School of Health Sciences, Hellenic Mediterranean University, Hellenic Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7414/10.01.2024
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Surgical Site Infection; Coronary Artery Bypass Grafting (CABG)
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group: Group A (No Intervention): No education and implementation of teleinterventions, whereas implementation of standard care based on the existing protocol of the Clinical Department is going to be applied
- Group B: nurse-led education (Experimental): The participants in Group B will be guided and trained by the principal investigator based on a specially designed educational booklet. Group B will also receive teleinterventions.
  Interventions: Other: Group B: nurse-led education
- Group C: nurse-led education and implementation of teleinterventions (Experimental): The participants in Group C will be guided and trained by the principal investigator based on a specially designed educational booklet. Group C will also receive teleinterventions and a guidance video will be presented to them
  Interventions: Other: Group C: nurse-led education and implementation of teleinterventions

INTERVENTIONS:
Other: Group B: nurse-led education — Group B: nurse-led education No educational video, will be shown to this group of patients
  Arms: Group B: nurse-led education
Other: Group C: nurse-led education and implementation of teleinterventions — Group C: nurse-led education and implementation of teleinterventions An educational video, made for the purposes of the study only, will be shown to them. This is the difference between the two groups
  Arms: Group C: nurse-led education and implementation of teleinterventions

SUMMARY:
The goal of this clinical trial is to determine if nurse-led education and tele-interventions can reduce the incidence of surgical wound infections in patients after coronary artery bypass surgery. The main questions it aims to answer are:

* Can nurse-led education reduce the rate of surgical wound infections after coronary artery bypass surgery?
* Does the addition of tele-interventions further decrease the incidence of these infections compared to standard care?

Researchers will compare three groups:

* Group A: Standard postoperative care
* Group B: Nurse-led patient education
* Group C: Nurse-led patient education plus tele-interventions

Participants will:

* Receive standard care, nurse-led education, or nurse-led education with tele-interventions
* Having regular follow-up as per group assignment
* Monitor and report infection during the study period

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who have undergone CABG with median sternotomy
* Proficiency in reading and writing in Greek
* Patients who provide written informed consent for participation in the study
* Patients who have access to a mobile phone and know how to use it
* Patients without difficulties in vision, speech, or hearing
* Patients at intermediate or high risk for developing surgical site infections, based on their scores in the risk stratification models described below

Exclusion Criteria:

* History of psychiatric illness, recent history of alcohol and/or substance abuse, dementia, and Alzheimer's disease
* Presence of an active infection within 2 weeks prior to the surgical procedure
* Preoperative hospitalization > 2 days
* Concurrent surgery on the aorta or heart valves
* Urgent or emergency nature of the surgical procedure
* Re-sternotomy aimed at surgical re-exploration of bleeding or implementation of cardiopulmonary resuscitation (CPR) in cases of cardiac arrest
* Patients in whom the sternum has not been closed after the completion of the surgical procedure and who are transferred to the cardiothoracic unit without sternum closure
* Active endocarditis
* Life expectancy < 6 months
* Lack of a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
nurse-led education and nursing teleinterventions on reducing the incidence of surgical site infections (SSIs) in patients who underwent planned coronary artery bypass grafting (CABG). | six months
  To investigate the effect of nurse-led education and the implementation of systematic nursing teleinterventions on reducing the incidence of surgical site infections (SSIs) in patients who underwent planned coronary artery bypass grafting (CABG).

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Mediterranean University, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No